CLINICAL TRIAL: NCT02941965
Title: Preimplantation Genetic Screening in Patients With Male Factor Infertility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Peace Maternity and Child Health Hospital (Other)
Responsible Party: Principal Investigator, He-Feng Huang, President, International Peace Maternity and Child Health Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPMCH2016001
Record Dates: First submitted 2016-10-19; First posted 2016-10-21 (Estimated); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Infertility, Male; Diagnosis, Preimplantation
MeSH Terms: conditions — Infertility, Male; Disease | interventions — Sperm Injections, Intracytoplasmic; Phosphatidylglycerols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICSI without PGS (Experimental): Selection of embryos are based on blastocyst morphology criteria on day 5. A maximum of 2 embryos will be transferred for each treatment cycle.
  Interventions: Procedure: ICSI without PGS
- ICSI with PGS (Experimental): PGS will be applied to select embryos on day 5, only euploid embryos will be transferred.
  A maximum of 2 embryos will be transferred for each treatment cycle.
  Interventions: Procedure: ICSI with PGS

INTERVENTIONS:
Procedure: ICSI without PGS — Selection of embryos are based on morphology criteria on the 5th day of ICSI.
  Arms: ICSI without PGS
Procedure: ICSI with PGS — PGS will be applied to selected embryos on the 5th day of ICSI.
  Arms: ICSI with PGS

SUMMARY:
This will be a prospective, randomized (1:1 ratio) clinical trial for patients with severe male-factor infertility with or without preimplantation genetic screening (PGS). Qualified 450 patients are randomized into either of two groups: group A will undergo intracytoplasmic sperm injection (ICSI) without PGS (225 cases), Group B will undergo ICSI with PGS (225 cases). The partners of all participants will receive the same protocol for ovarian stimulation and standardized luteal phase support.

The target population will be patients with severe male-factor infertility aged between 20 and 55 years, diagnosed by the ESHER Criteria (Non-obstructive oligospermia，asthenspermia). Women with other reasons of infertility (eg. advanced age, anovulation, endometriosis, and premature ovarian failure) are excluded.

The randomization will take place 3-6 days after the oocyte pick-up day by a computer randomization system. The pregnancy test results, pregnancy complications, congenital anomalies, neonatal complications will be followed up by checking medical records and telephone calls.

ELIGIBILITY:
Inclusion criteria

1. Male partner age of 20-55 years old, Chinese.
2. Male partner has severe male infertility (defined as a semen concentrate less than 5×10^6/ml, and/or with a progressive motility less than 10%).
3. Proposed ICSI to assist pregnancy.
4. Fully explain the nature of the research and obtain the informed consent of the subject before carrying out any procedure in the research protocol. If a subject is not capable of expressing opinions, the legal representative of the subject can sign the informed consent on behalf of the subject.

Exclusion criteria

Any one of the following criteria should be excluded from this study:

1. Male partner had been diagnosed with obstructive azoospermia, sexual dysfunction, and immune infertility.
2. Female partner at 38 years of ages and older.
3. Female partner has uterine abnormalities such as uterine malformations (unicornuate uterus, mediastinal uterus, double uterus, double horn uterus, etc.), adenomyosis, submucosal fibroids or intrauterine adhesions.
4. Female partner has a history of recurrent abortion, including biochemical pregnancy (≥3 time miscarriages).
5. One of the couples has abnormal chromosomal karyotypes, excluding chromosomal polymorphisms.
6. Female partner has contraindications for assisted reproduction, such as poorly controlled type I or type II diabetes mellitus; undiagnosed liver disease or abnormal liver function (abnormal serum liver enzymes); kidney disease or abnormal kidney function; severe anemia; history of deep venous thrombosis; history of pulmonary embolism; history of cerebrovascular accident; poorly controlled hypertension or diagnosed heart disease; history of cervical cancer, endometrial cancer or breast cancer; unexplained vaginal bleeding.
7. Male partner has contraindications for assisted reproduction, such as poorly controlled type I or type II diabetes mellitus; undiagnosed liver disease or abnormal liver function (abnormal serum liver enzymes); kidney disease or abnormal kidney function; severe anemia; history of deep venous thrombosis; history of pulmonary embolism; history of cerebrovascular accident; poorly controlled hypertension or diagnosed heart disease.
8. One of the couple refuses to cooperate with the study.
9. Patients who have been included in the experimental group or control group of this study.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2017-07-18 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
live birth rate | 42 weeks
  This will be based on the outcome of either the PGS+ICSI or the outcome of the ICSI after first embryo transfer cycle.

SECONDARY OUTCOMES:
clinical pregnancy rate | 35 days after embryo transfer
  Clinical pregnancy was defined as an observation of gestational sac via ultrasonography.
implantation rate | 11-12 weeks after embryo transfer
  Implantation rate was defined as the percentage of fetal heart beat among total transferred embryos at 12 weeks' gestational age.
biochemical pregnancy rate | 2 weeks after embryo transfer
  Biochemical pregnancy was defined as numbers of women with an elevated serum β-hCG level of more than 10 mIU/ml.
pregnancy loss rate | 28 gestational weeks in maximum
  Pregnancy loss is defined as any reason that resulted in failure of an embryo to develop, embryonic or fetal death, or spontaneous expulsion of a pregnancy.
ectopic pregnancy rate | 12 gestational weeks in maximum
  Ectopic pregnancy is defined as an embryo implanted outside the uterine.
Congenital Anomalies rate | 1 day after delivery
  Congenital anomaly included deformity and development abnormality of any organs or systems.
neonatal complication rate | 1 day after delivery
  Neonatal complication includes neonatal respiratory disorders, neonatal cerebral palsy, neonatal encephalopathy and other disease that should been sent into neonatal ICU.

CONTACTS AND LOCATIONS:
Overall Officials: He-Feng Huang, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- International Peace Maternity & Child Health Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin X, Wu D, Zhang C, Wang L, Lu Y, Zhou P, Zhou C, Jin L, Wang L, Zhu H, Pan J, Xu C, Chen S, Gao L, Li L, Zhang S, Wu Y, Sun Y, Mol BW, Huang H. Preimplantation genetic testing for aneuploidy versus no genetic testing in couples undergoing intracytoplasmic sperm injection for severe male infertility: multicentre, open label, randomised controlled trial. BMJ. 2025 Dec 23;391:e084050. doi: 10.1136/bmj-2025-084050. PMID 41436190
- [Derived] Lin XH, Guo MX, Wu DD, Lu Y, Zhang JL, Zhou CL, Jin L, Wang L, Zhang C, Xu CM, Chen SC, Zhang SY, Sun XX, Wu YT, Sun Y, Huang HF. Preimplantation genetic testing for aneuploidy in severe male factor infertility: protocol for a multicenter randomised controlled trial. BMJ Open. 2022 Jul 13;12(7):e063030. doi: 10.1136/bmjopen-2022-063030. PMID 35831058
- [Derived] Cornelisse S, Zagers M, Kostova E, Fleischer K, van Wely M, Mastenbroek S. Preimplantation genetic testing for aneuploidies (abnormal number of chromosomes) in in vitro fertilisation. Cochrane Database Syst Rev. 2020 Sep 8;9(9):CD005291. doi: 10.1002/14651858.CD005291.pub3. PMID 32898291